CLINICAL TRIAL: NCT06335615
Title: Examining the Effectiveness, Mediators, and Moderators of a Brief Acceptance Intervention for Stress to Improve Students' Well-Being: A Randomized Controlled Trial
Brief Title: A Brief Acceptance Intervention for Stress to Improve Students' Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Jaap Lancee, Assistant Professor, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMG-5790_2023
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Stress
Keywords: Acceptance; Acceptance and Commitment Therapy; Brief Intervention; Student Mental Health

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group follows a one-hour in-person intervention focused on acceptance of stress. Each participant follows this intervention individually.
  Interventions: Behavioral: Brief Acceptance Intervention
- Control (Active Comparator): The control group follows a 20-minute online psychoeducation at home. Each participant follows this intervention individually.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Brief Acceptance Intervention — The intervention consist of explanations and exercises about acceptance of stress. The intervention starts with a welcome, after which participants do jumping jacks and then breath through a straw to induce an uncomfortable experience. Next, a Chinese finger trap is used to show the automatic, but often not useful, reaction to avoid stress. Participants then watch a short video that introduces the concept of acceptance, and they do a short, guided meditation. Afterwards, they do the straw exercise again, but this time with instruction to examine and allow uncomfortable experiences. The session ends with a recap and the introduction of the home exercise. Participants install an app that reminds them every hour to do a three-second meditation in which they pay attention to their breathing and body in an accepting way.
  Arms: Intervention
Behavioral: Psychoeducation — In the psychoeducation, participants learn about the stress response, mindfulness, and acceptance. For this, they are guided through a vignette about a student who struggles with stress and then develops a more accepting stance towards it. The psychoeducation explains how acceptance can help to deal with stress but does not instruct participants to apply this in their own life.
  Arms: Control

SUMMARY:
The goal of this randomized controlled trial is to test a brief psychological intervention that focusses on acceptance of stress in a student population. The main questions it aims to answer are:

* Does this brief acceptance intervention increase the well-being of students in the short term?
* By which mechanisms does this effect occur?
* What are moderating factors of this effect?

Half of the participants follow a one-hour intervention, which includes

* psychoeducation and metaphors about stress and how acceptance can help to deal with it
* experiential exercises
* mindfulness meditation
* mindfulness homework practice

Students that receive the intervention will be compared to students that merely received psychoeducation about stress and acceptance to see if the intervention lead to larger increases in well-being.

ELIGIBILITY:
Inclusion Criteria:

* Student at the University of Amsterdam in the Bachelor's programme psychology or communication science

Exclusion Criteria:

* Panic Disorder as measured with the Rapid Measurement Toolkit-20 (Batterham et al., 2020; cutoff at 9)
* Asthma, Chronic Obstructive Pulmonary Disease (COPD), another lung disease (including covid-related lung complaints), or tightness of chest
* Pregnancy
* Physical disability that limits ability to move and jump

Ages: 17 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Psychological Well-Being | Change from baseline (1 - 14 days before the intervention/psychoeducation) to post measurement (3 days after the intervention/psychoeducation)
  Psychological well-being was measured with the General Health Questionnaire-12 (GHQ-12, Goldberg & Williams, 1988), which is a unidimensional measure of mental health with good psychometric properties (Romppel et al., 2013). Higher scores on the GHQ-12 indicate more psychological distress and lower well-being.

SECONDARY OUTCOMES:
State Anxiety | Change from baseline (1 - 14 days before the intervention/psychoeducation) to post measurement (3 days after the intervention/psychoeducation)
  The six-item version of the Spielberger State-Trait Anxiety Inventory (STAI; Marteau & Bekker, 1992) is a brief, valid, and reliable questionnaire to assess participants' state anxiety.
Study Stress | Change from baseline (1 - 14 days before the intervention/psychoeducation) to post measurement (3 days after the intervention/psychoeducation)
  A single question was used for study-related stress: How much stress related to studying are you currently experiencing on a scale of 0 (no stress) to 10 (extreme stress)?
Interoceptive awareness | Change from baseline (1 - 14 days before the intervention/psychoeducation) to post measurement (3 days after the intervention/psychoeducation)
  The Multidimensional Assessment of Interoceptive Awareness (MAIA-2, Mehling et al., 2018) measured body awareness. In line with Ferentzi and colleagues (2020) and for enhanced psychometric validity, we will combine six subscales to measure a general level of interoception.
Psychological Flexibility | Change from baseline (1 - 14 days before the intervention/psychoeducation) to post measurement (3 days after the intervention/psychoeducation)
  The Comprehensive Assessment of Acceptance and Commitment Therapy Processes questionnaire (CompACT; Francis et al., 2016) measures the underlying processes of Acceptance and Commitment Therapy. It has good psychometric properties (Francis et al., 2016). We will be especially interested in the subscale openness to experience, which corresponds to the processes of acceptance and defusion.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All anonymized individual participant data will be shared. Demographic information that may lead to identification of individuals, such as open questions about education and gender will be removed.
Supporting Information: ICF, Analytic Code
Time Frame: Data will be made available with publication of the journal article. There is no specified time limit for availability.